CLINICAL TRIAL: NCT03883321
Title: Interest of Cognitive-behavioral Therapies Based on the CBSM (Cognitive Behavior Stress Management) for the Management of Patients Suffering From Pain Related to Cancer.
Brief Title: EssaiClinique_CBSM
Acronym: CBSM
Status: Terminated | Type: Observational
Why Stopped: few patient feedback and principal investigator disponibility
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC17.291; 2017-A02618-45 (Other: ID RCB)
Record Dates: First submitted 2019-01-15; First posted 2019-03-20 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Perceived Stress
Keywords: stress management; CBSM; Chronic Pain; Cancer
MeSH Terms: conditions — Chronic Pain; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CBSM: Patients included in this group participate in the CBSM program. They attend 10 sessions of stress management according to the CBSM program, 9 take place over 3 months and the tenth session takes place 3 months after the 9th session. The session is composed of relaxation and cognitive and behavioral therapy, which is carried out in groups of 8 to 10 patients
  Interventions: Other: Cognitive behavioral stress management
- Waiting list: The CBSM group is compared to the "waiting list" group that does not benefit from the CBSM program. After completing their assessment in the "waiting list" group, patients in this group will be integrated into the CBSM group but will not be evaluated as such.

INTERVENTIONS:
Other: Cognitive behavioral stress management — Management of patients in 10 group sessions with cognitive and behavioral therapies associated with relaxation in order to learn how to manage stress
  Groups: CBSM

SUMMARY:
The CBSM is a program combining cognitive and behavioral therapies, relaxation provided in groups of 8 to 10 patients. This program has demonstrated benefits in stress management skills, adaptive strategies, anxiety, quality of life, social inclusion, medication adherence, depression, therapeutic alliance, and general well-being. It would also improve breast cancer survival after adjuvant therapy. This program has been put in place at the center of pain for patients with cancer pain in any stage. This study aims to evaluate the benefits of this technique on a patient population suffering from chronic pain related to cancer.

DETAILED DESCRIPTION:
Methodology: Observational study, prospective, open, mono-centric, comparative, evaluating a psychosocial intervention type CBSM versus no intervention (group "waiting list").

Main Objective: To evaluate the impact of the implementation of a "CBSM" program on the stress management capacities of a pilot group of 30 patients followed at the pain center of Grenoble-Alpes University Hospital for chronic pain related to cancer or its treatment, compared to a control group "waiting list"

Primary Outcome: Measurement of emotional stress (PSS14)

Secondary objective:

Determine patients' interest in this program and the feasibility of the program.

Determine patient satisfaction with this program To evaluate the impact of the program on the quality of life of patients. To evaluate the impact of the program on the handicap perceived by the patients in connection with their pains.

Evaluation of the impact of the program on the pain of the patients (on the daily behavior).

Evaluation of the impact of the program on depression and anxiety. Determine the impact of the 3-month program of the 9th session on the different dimensions described above

Inclusion criterion:

* Over 18,
* Currently treated or treated for cancer (solid or otherwise), any stage combined.
* With chronic pain related to cancer or its treatment
* Never benefited from the management of stress by this technique
* Knowing how to read, write and speak French
* Person affiliated with social security or beneficiary of an equivalent plan.

Criteria of non-inclusion:

* Life expectancy of less than 6 months
* Patients unable to travel for 10 sessions on the structure (CHUGA)
* Person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure.

Number of patients included: a minimum of 30 patients including, a minimum of 15 in the CBSM group and a minimum of 15 in the "waiting list" group (patients included in the waiting list group will participate in the CBSM program but will not be not analyzed in the CBSM group)

ELIGIBILITY:
Inclusion Criteria:

* Over 18,
* Currently treated or treated for cancer (solid or otherwise), any stage combined.
* With chronic pain related to cancer or its treatment
* Never benefited from the management of stress by this technique
* Knowing how to read, write and speak French
* Person affiliated with social security or beneficiary of an equivalent plan.

Exclusion Criteria:

* Life expectancy of less than 6 months
* Patients unable to travel for 10 sessions on the structure
* Person deprived of liberty by judicial or administrative decision, person subject to a legal protection measure.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient being treated for cancer, undergoing treatment or having completed treatment, at any stage and suffering from chronic pain
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Measurement of emotional stress (PSS14) | evaluation at the beginning of the meeting and at 9 weeks
  assessment of the evolution of stress over a period of 3 months: Questionnaire PSS14

SECONDARY OUTCOMES:
Inclusion rate | up to 18 months
  ratio of number of patients who agreed to participate in the program to the number of patients to whom the program was proposed
Satisfaction | at 6 months
  Satisfaction rate of CBSM program with a questionnaire
Measurement of quality of life | evaluation at the beginning of the meeting and at 9 weeks and then at 3 months
  Evaluate the impact of the program on the quality of life of patients with a Physical and Mental Health Summary Scales with 12 questions (SF12) questionnaire
Pain Disability Index (PDI) | evaluation at the beginning of the meeting and at 9 weeks and then at 3 months
  Evaluate the impact of the program on disability perceived by patients in relation to their pain: PDI questionnaire
concise questionnaire on pain short version (QCD) | evaluation at the beginning of the meeting and at 9 weeks and then at 3 months
  Evaluation of the impact of the program on patients' pain (on daily behavior) with QCD questionnaire
Hospital Anxiety and Depression Scale (HADS) | evaluation at the beginning of the meeting and at 9 weeks and then at 3 months
  Evaluation of the impact of the program on depression and anxiety with HADS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Claudine BERTHOZAT, MD, Principal Investigator — pain center, Grenoble University Hospital
Locations (1):
- Grenoble University Hospital, La Tronche, Isère, France

IPD SHARING:
Plan to Share IPD: Undecided